CLINICAL TRIAL: NCT01529463
Title: Effect of Post Discharge Follow-up on Readmission Rates for Congestive Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Other Study IDs: 11-01-001-E
Record Dates: First submitted 2011-01-25; First posted 2012-02-08 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2012-12

CONDITIONS: Congestive Heart Failure; Systolic Dysfunction
Keywords: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Disease Management

SUMMARY:
The purpose of this study is to test the hypothesis that a comprehensive post-discharge disease management system is more effective in reducing the readmission rate for heart failure patients compared to standard care.

DETAILED DESCRIPTION:
Heart failure, a disease that affects a large proportion of the aging population, continues to be associated with poor outcomes especially in patients who require hospitalization. Each year, nearly 1 million Americans are newly diagnosed with congestive heart failure and currently, there are at least 5 million Americans living with this chronic disease. The number of patients with heart failure is expected to reach 10 million by the year 2037.This population consumes a large proportion of health care resources with the main cost being hospitalization. The heart failure 30-day readmission rates hover around 25% nationally, with an approximate cost of $7,000 per hospitalization.

In an effort to improve care and reduce costs, heart failure disease management programs are becoming more prevalent. Recent data suggests that multi-disciplinary disease management programs may reduce mortality and hospitalizations as well as improve costs, patients' ability to self-care, and quality of life. It provides a means to increase the use of evidence-based therapies, improve patient education, and decrease resource usage. Heart failure management programs involve early assessment, optimized treatment, easy access to care, and education and psychosocial support.

Patients hospitalized for decompensated congestive heart failure are among the highest risk group for morbidity and mortality among people with chronic heart failure and a large proportion of this risk occurs early after discharge. Thus, the goals of these programs should include managing the gap between the inpatient and outpatient settings and should ideally involve a multidisciplinary team in order to serve these patients in a comprehensive manner. We propose to determine the relative efficacy of a post-discharge disease management system.

PRIMARY OBJECTIVE:

The primary objective of this study is to determine if the time to first hospital readmission can be lengthened using a disease management model.

STUDY DESIGN:

This is a prospective, one year pilot study that will enroll patients admitted to Saint Francis Hospital and Medical Center (SFHMC) with the admitting diagnosis of acute decompensated heart failure that have been referred to the Congestive Heart Failure Disease(CHF)Management Program by the attending physician. The patients will be enrolled in the study and followed for a maximum of 90 days post-discharge. A case control group of 60-100 subjects will also be established for primary endpoint analysis.

METHODS:

Patients who meet study criteria, informed consent will be obtained before hospital discharge or at the first Disease Management visit. Patients will be followed for 90 days post-discharge. Clinic visits, homecare agency and visits, heart failure education class attendance, and dates of hospital readmission will be tracked. Descriptive characteristics of patients will be recorded at the time of enrollment. Descriptive characteristics include demographics, etiology of heart failure, symptoms, physical assessment, current medications, lab results, and diagnostic test results.

In everyday practice, the Congestive Heart Failure Disease Management Program administers clinical questionnaires to patients to assess quality of life and heart failure management knowledge. The clinical questionnaires that constitute standard of care for these patients include:

* Atlanta Heart Failure Knowledge Test: given to each patient at the first Disease Management visit and after attending the Congestive Heart Failure educational series to determine level of understanding of self-management of heart failure.
* Kansas City Living with Cardiomyopathy Questionnaire (KCCQ): This is a validated quality of life survey. The questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality. This survey is administered to each patient upon enrollment into the Disease Management Program and prior to discharge from the Disease Management Program.

Results from these questionnaires will be collected and enrollment and discharge scores will be compared for improvement in level of understanding of self-management of heart failure and overall quality of life.

One hundred consecutive patients discharged from SFHMC with a primary diagnosis of acute decompensated heart failure that have not been referred to the Congestive heart Failure Disease Management Program will undergo retrospective chart review to establish a case control group. The study team will perform a retrospective chart review to abstract the following data: hospital admission date, hospital discharge date, attending physician, age, and ejection fraction.

RISKS AND SAFETY:

There are no physical or psychological risks associated with this study. The study does not involve any experimental treatments or invasive therapies. There is a less than minimal risk of disclosure of clinical information maintained in the file linking the patient's medical record to the data. This file will be kept to allow follow up tracking for heart failure re-admission. The file will be password protected and available solely to the site Principal Investigator and Institutional Review Board-approved study staff. At the end of the study, following data analysis and publication of an abstract and paper in appropriate peer reviewed journal(s), the file linking the patient names to the case report forms will be destroyed.

POTENTIAL BENEFITS:

There are no potential benefits to patients whose records are entered into the database. The potential benefit is to society and future patients diagnosed with heart failure. Implementation of a disease management model may improve functional and clinical outcomes through more productive interactions between patients and providers. A disease management model may decrease hospital re-admission rates and the associated cost. If this disease management model proves effective, the results will provide a framework for expanding care opportunities and for establishing a new model for heart failure patients in this health care system as well as in other systems.

DATA ANALYSIS:

The primary endpoint will be assessed as a continuous variable using Kaplan Meier survival analysis. The time to all-cause readmission and readmission for heart failure will be assessed using this methodology. The time to all-cause readmission and readmission for heart failure in the CHF Disease Management Group will be compared to aggregate hospital readmission data.

The QOL questionnaire will be analyzed using a t-test comparing enrollment and 2 month KCCQ scores. The validity of each individual domain of this questionnaire has been independently established and all components of the summary score are considered valid representations of their intended domains.

ELIGIBILITY:
Inclusion Criteria:

* Age =/or >18
* Admitted to the Heart Failure Unit with acute decompensated heart failure
* Referred to the Congestive Heart Failure Disease Management Program

Exclusion Criteria:

* Age<18
* Mentally incapacitated
* Discharge to a skilled nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with an admitting diagnosis of acute decompensated heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The time from hospital discharge to first hospital readmission or death. | basline and 1 month
  The primary endpoint will be assessed as a continuous variable. Survival curves will be produced using Kaplan-Meier analysis for both the CHF Disease Management Group and the case control group. A Cox regression-based test will be used to test differences in survival between the CHF Disease Management Group and the case control group. If case control subjects cannot be exactly matched on covariates to CHF Disease Management subjects, inverse probability of treatment weights (obtained via logistic regression) will be applied to correct for covariate imbalances between the two groups.

SECONDARY OUTCOMES:
The time from hospital discharge to unplanned hospital admission for acute decompensated heart failure. | baseline and 3 months
  3 months minus baseline
Change in quality of life. | baseline and 2 months
  Kansas City Living with Cardiomyopathy Questionnaire will be analyzed using a paired t-test comparing baseline and 2 month scores.
Mean readmission cost for each patient for total cost for each readmission. | baseline and 3 months
  Average costs for the medical management group versus the disease management group will be calculated.
Improvement in knowledge of Heart Failure | baseline and 2 months
  Atlanta Heart Failure Knowledge Test baseline score minus 2 month score

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Soucier, M.D., Principal Investigator — Saint Francis Hosptial and Medical Center
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States